CLINICAL TRIAL: NCT07205900
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate Efficacy, Safety, and Tolerability of HM15275 for 36 Weeks in Obese or Overweight Subjects Without Diabetes Mellitus
Brief Title: Study to Evaluate HM15275 in Obese or Overweight Subjects Without Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-OBCT-201
Record Dates: First submitted 2025-09-16; First posted 2025-10-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Obese; Obesity
Keywords: Obese; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomly assigned in a 1:1:1:1:1 ratio to 1 of the 5 treatment arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment assignment will remain blinded to participants, investigators/study personnel, and sponsor's study team conducting the study. Participants who meet all criteria for enrollment will be centrally assigned randomized to study drug using an Interactive Web Response System (IWRS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HM15275 (Experimental): Participants will receive HM15275 via subcutaneous (SC) injection.
  Interventions: Drug: HM15275
- Placebo of HM15275 (Placebo Comparator): Participants will receive placebo of HM15275 via subcutaneous (SC) injection.
  Interventions: Drug: Placebo of HM15275

INTERVENTIONS:
Drug: HM15275 — HM15275 is a sterile solution for subcutaneous injection, supplied pre-filled syringes.
  Arms: HM15275
Drug: Placebo of HM15275 — A sterile, matching solution supplied in pre-filled syringes.
  Arms: Placebo of HM15275

SUMMARY:
This Study is a Phase 2 Study to Evaluate Efficacy, Safety, and Tolerability of HM15275 for 36 Weeks in Obese or Overweight Subjects Without Diabetes Mellitus.

DETAILED DESCRIPTION:
HM-OBCT-201 is a Phase 2, randomized, double-blind, placebo-controlled, multicenter, parallel group study designed to evaluate the efficacy, safety, and tolerability of HM15275 treatment over 36 weeks in obese or overweight adults without Type 2 diabetes mellitus (T2DM).

The study will enroll adult participants with obesity (body mass index [BMI] ≥30 kg/m2 and ≤50 kg/m2) or with overweight (BMI ≥27 kg/m2 and <30 kg/m2) with at least 1 weight-related comorbidity. Patients with T2DM will be excluded.

Participants in this study will be randomly assigned in a 1:1:1:1:1 ratio to 1 of the 5 treatment arms. Randomization will be stratified by sex (female vs male) and BMI (<35 vs ≥35 kg/m2).

All participants will undergo a 6-week screening period, a 36-week treatment period (including the dose-titration phase with weekly subcutaneous [SC] injection), and a 4-week safety follow-up period.

ELIGIBILITY:
Key Inclusion Criteria

1. Participant's age at the time of signing the informed consent:

   * United States: 18 to 75 years (inclusive)
   * Korea: 19 to 75 years (inclusive)
2. BMI ≥30 kg/m² and ≤50 kg/m², or ≥27 kg/m² and <30 kg/m² with ≥1 weight-related comorbidity
3. Body weight change <5% over the past 3 months prior to screening
4. Capable of giving signed informed consent, ability and willingness to comply with all protocol procedures

Key Exclusion Criteria:

1. Type 1 diabetes mellitus or T2DM, or HbA1c ≥6.5% / FPG ≥126 mg/dL
2. Obesity due to endocrine/genetic disorders
3. Planned or prior obesity surgery (unless >1 year ago for liposuction/abdominoplasty), or device-based obesity therapy (unless removed >6 months ago)
4. Personal history or current diagnosis of acute or chronic pancreatitis or factors that may increase the risk of pancreatitis, such as a history of cholelithiasis (without cholecystectomy) or alcohol abuse.
5. Personal or family history of medullary thyroid carcinoma (MTC) or a known genetic condition (e.g., multiple endocrine neoplasia type 2) that predisposes the participant to MTC.
6. Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
7. History or current diagnosis of congestive heart failure (NYHA class Ⅲ or Ⅳ), or myocardial infarction, stroke, unstable angina, transient ischemic attack, or revascularization procedure (e.g., stent or bypass graft surgery) within 3 months prior to screening visit
8. Personal history or current diagnosis of acute or chronic pancreatitis or factors that may increase the risk of pancreatitis, such as a history of cholelithiasis (without cholecystectomy) or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight. | Up to 41 weeks
  Percent change in body weight from Week 1 to Week 37, measured using a standardized, calibrated scale under fasting conditions.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 41 weeks
  Number of participants with adverse events (AEs) after multiple subcutaneous (SC) doses.

OTHER OUTCOMES:
Plasma concentration profile | Up to 41 weeks
  Plasma concentration profile of HM15275 after multiple subcutaneous (SC) doses.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - ProSciento Inc, Chula Vista, California
  - Accellacare of Duly - Duly Oak Lawn, Oak Lawn, Illinois
  - Accellacare of McFarland, Ames, Iowa
  - Accellacare of Cary - Cary Medical Group, Cary, North Carolina
  - Accellacare of Hickory, Hickory, North Carolina
  - Raleigh Medical Group, P.A., Raleigh, North Carolina
  - Accellacare of Piedmont - Piedmont HealthCare, Statesville, North Carolina
  - Accellacare of Wilmington, LLC, Wilmington, North Carolina
  - Accellacare of Winston Salem, Winston-Salem, North Carolina
  - Accellacare of Charleston, Mt. Pleasant, South Carolina
  - Accellacare of Bristol-PAC of Tennessee, Bristol, Tennessee
  - Bristol-Internal Medicine and Pediatric Associates of Bristol, P.C., Bristol, Tennessee
  - Velocity Clinical Research, Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No